CLINICAL TRIAL: NCT01540305
Title: A Randomized Double-blind Trial of Repetitive Transcranial Magnetic Stimulation in Obsessive -Compulsive Disorder With Three Months Follow-up
Brief Title: Efficacy Study of Transcranial Magnetic Stimulation for Treatment of Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Joaquim Brasil-Neto, Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49/09
Record Dates: First submitted 2012-02-15; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Transcranial Magnetic Stimulation; Treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Magnetic Stimulation (Active Comparator): Actual transcranial magnetic stimulation of supplementary motor areas bilaterally.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham transcranial magnetic stimulation over the supplementary motor areas.
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS was administered by means of a NEURO-MS (NEUROSOFT LTD®, Russia) with a focal 8-shaped 70 mm coil. Stimulation parameters were 1-Hz, 20-min trains (1200 pulses/day) at 100% of resting MT, once a day, 5 days a week, for 2 weeks.
  Other Names: Neuro-MS Transcranial Magnetic Stimulator
  Arms: Transcranial Magnetic Stimulation
Device: Sham repetitive transcranial magnetic stimulation — The sham treatment was performed using the Neurosoft ® sham coil. A metal plate placed inside this coil prevents the magnetic field from stimulating the cortex. This coil looks and sounds like an active coil.
  Other Names: Neurosoft sham coil
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
This study aimed at verifying whether sessions of repetitive transcranial magnetic stimulation over a certain brain area (the supplementary motor area) could be useful in the relief of Obsessive-Compulsive Disorder symptoms.

DETAILED DESCRIPTION:
Patients were randomly administered either real (n = 12) or sham (n = 10) rTMS, once a day, 5 days a week, for 2 weeks. Randomization was performed according to a computer-generated schedule. Subjects and scale-rater physician were blind to treatment status of individuals. Only the rTMS administrator was aware of group allocations. Treatment response was assessed by self-and clinician-rated scales before treatment, immediately after treatment and 3 months thereafter, with the same examiner following a subject throughout the study. All patients included in the study had failed adequate pharmacological treatment for at least 2 antiobsessional drugs. Their prescription drugs were continued without change in dosage regimens throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 60 years
* diagnosis of obsessive-compulsive disorder (OCD) according to DSM-IV-TR criteria and having OCD of at least moderate severity (YBOCS score of 16 or above).

Exclusion Criteria:

* subjects with comorbid psychiatric disorders (except depression - HAM-D ) or history of drug abuse
* significant head injury, or of any neurosurgical procedure
* pregnant women
* patients with metal implants or illnesses that prevent attendance to sessions
* patients with a history of seizure or bearing pacemakers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes in Y-BOCS scale scores relative to baseline | assessments were at baseline, at 2 weeks and at 3 months
  Y-BOCS: Yale-Brown Obsessive-Compulsive Scale

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Brasil-Neto, MD, PhD, Study Director — University of Brasilia
Locations (1):
- Laboratory of Neurosciences and Behavior, Biology Institute, University of Brasília, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Mantovani A, Simpson HB, Fallon BA, Rossi S, Lisanby SH. Randomized sham-controlled trial of repetitive transcranial magnetic stimulation in treatment-resistant obsessive-compulsive disorder. Int J Neuropsychopharmacol. 2010 Mar;13(2):217-27. doi: 10.1017/S1461145709990435. Epub 2009 Aug 20. PMID 19691873
- [Background] Mantovani A, Lisanby SH, Pieraccini F, Ulivelli M, Castrogiovanni P, Rossi S. Repetitive transcranial magnetic stimulation (rTMS) in the treatment of obsessive-compulsive disorder (OCD) and Tourette's syndrome (TS). Int J Neuropsychopharmacol. 2006 Feb;9(1):95-100. doi: 10.1017/S1461145705005729. Epub 2005 Jun 28. PMID 15982444